CLINICAL TRIAL: NCT06492538
Title: Biometric Changes After Intervention of Anterior Chamber Angle : an Observational Study
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xinbo Gao, associate professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2023KYPJ304
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Angle-closure Glaucoma; Minimally Invasive Glaucoma Surgery; Goniosynechialysis; Goniotomy; Glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- laser peripheral iridotomy/iridoplasty group: based on angle closure mechanism, procedures were chosen LPI alone or combined with ALPIp.
  LPI: laser peripheral iridotomy; ALPIp: argon laser peripheral iridoplasty.
  Interventions: Procedure: various types of angle interventions
- peripheral iridectomy based surgery combo: SPI combined with GSL or GSL+GT SPI: surgical peripheral iridectomy GSL:goniosynechialysis GT: goniotomy GSL and GT are both guided by surgical goniolens
  Interventions: Procedure: various types of angle interventions
- phacoemulsification and intraocular lens implantation based surgery combo: PEI: phacoemulsification and intraocular lens implantation surgery combo includes GSL alone or GSL+GT.
  Interventions: Procedure: various types of angle interventions
- ab interno goniotomy: GT was performed in the nasal-inferior quadrant or nasal quadrant because the collector channels were mainly concentrated in the nasal quadrant, by inserting the tip of a microblade (TMH; Tanito Microhook, Inami & Co., Ltd., Tokyo, Japan) into Schlemm's canal, and then the inner wall of Schlemm's canal and trabecular meshwork was incised over 120°
  Interventions: Procedure: various types of angle interventions
- Schlemm canaloplasty: performed in the nasal quadrant by the collector channels were mainly concentrated in the nasal quadrant, by inserting the tip of a microblade (TMH; Tanito Microhook, Inami & Co., Ltd., Tokyo, Japan) into Schlemm's canal, and then the inner wall of Schlemm's canal and trabecular meshwork was incised over 120°
  Interventions: Procedure: various types of angle interventions

INTERVENTIONS:
Procedure: various types of angle interventions — procedures include laser peripheral iridotomy (LPI) to relieve pupillary tissue and deepen peripheral anterior chamber depth, Argon laser peripheral iridoplasty (ALPIp) to stimulate iris contraction and widen the angle, and mechanical separation of adhered angle tissues using instruments like goniosynechialysis hooks or iris repositor. Ab interno goniotomy using instruments like retina hooks, trabeculectomy hooks, or cannulas are used to incise trabecular meshwork and Schlemm's canal walls to enhance aqueous humor outflow.

SUMMARY:
The drainage angle in the anterior chamber of the eye mediates the outflow of aqueous humor, and pathological changes here can lead to high intraocular pressure and glaucoma. Minimally invasive glaucoma surgery, particularly angle surgery, has advanced recently, allowing clear visualization of angle structures like the trabecular meshwork and Schlemm's canal using surgical goniolens. Techniques for angle intervention include widening the angle, reopening closed angles, and rebuilding outflow pathways using methods such as laser peripheral iridotomy, Argon laser peripheral iridoplasty, and mechanical separation of adhered tissues. Our research team plans to conduct imaging studies to track the healing of angle tissues post-surgery, aiming to support innovation and standardization of minimally invasive angle surgery.

DETAILED DESCRIPTION:
Pathological elevated intraocular pressure is one of the most important disease characteristics of glaucoma. Blockage of aqueous humor outflow within the eye is the primary cause of high intraocular pressure. The drainage angle in the anterior chamber of the eye mediates the outflow of aqueous humor. Pathological changes in this area can lead to the development of high intraocular pressure and glaucoma, such as primary angle closure glaucoma (PACG) caused by angle closure. Minimally invasive glaucoma surgery has rapidly developed in recent years, with angle surgery being a major branch. With the use of surgical goniolens, structures within the angle, such as trabecular meshwork and Schlemm's canal, can be visualized clearly during surgery. Methods for angle intervention include but not limit ed to widening the peripheral anterior chamber angle, reopening adhered or appositionally closed angles, and rebuilt outflow pathways by incising diseased areas to increase aqueous humor outflow. Techniques include laser peripheral iridotomy (LPI) to relieve pupillary block and deepen the peripheral anterior chamber, Argon laser peripheral iridoplasty (ALPIP) to stimulate iris contraction and widen the angle, and mechanical separation of adhered angle tissues using instruments like goniosynechialysis hooks or iris repositors. Surgical incision using instruments such as Microhook, trabeculectomy hooks, or cannulas can be performed to remove the diseased inner wall of Schlemm's canal and the diseased trabecular meshwork either partially or circumferentially. However, the healing and outcomes of angle tissues following invasive angle interventions, and their impact on surgical outcomes, remain unclear. Therefore, our research team proposes to conduct imaging observation studies to track, observe, and quantify the status of the angle, exploring the healing process of angle tissues. This aims to provide theoretical support for the innovation and standardization of minimally invasive angle surgery.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma patients eligible for standalone or combined angle intervention surgeries, such as LPI, LPIP, goniosynechialysis, trabeculotomy alone or combined with surgical iridectomy or phacoemulsification and intraocular lens implantation;
* Patients capable of undergoing preoperative examinations including CASIA2-OCT (anterior segment OCT), UBM, slit-lamp gonioscopy, IOL Master (or other optical biometry);
* Patients willing to participate in this study, signing informed consent, and agreeing to follow-up according to the study protocol.

Exclusion Criteria:

* Patients with severe ocular conditions such as corneal infection, ulcer, trauma, ocular tumors, retinal vascular occlusion, and retinal detachment;
* Those with various types of eye diseases that affect ocular parameter acquisition or interfere with visual field examination;
* Long-term local or systemic use of glucocorticoids;
* Patients with severe systemic diseases;
* Pregnant or lactating women;
* Unable to complete 12-month postoperative follow-up.

Ages: 30 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with glaucoma typically present with: IOP > 21 mmHg with or without the use of ocular hypotensive medications; (3) with obvious glaucomatous optic neuropathy [cup-to-disc (C/D) ratio ≥ 0.7, C/D ratio asymmetry > 0.2, or rim width at the superotemporal and inferotemporal < 0.1 vertical diameter of the optic disc], and glaucomatous visual field defects, such as nasal step, arcuate scotoma, and paracentral scotoma;
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in biological parameters of the anterior chamber angle | 12 months
  Biological parameter changes in the anterior chamber following angle intervention surgery will be measured using Casia2-OCT

SECONDARY OUTCOMES:
success rate of angle intervention surgeries | 12 months
  complete success was defined as postoperative IOP within the range of 6-18 mmHg, and a reduction of 20% from baseline without loss of light perception, additional ocular hypotensive medication, and reoperation. The definition of qualified success was similar to that of complete success, except for the need for ocular hypotensive medications. Postoperative ocular hypotensive medications were adjusted according to the IOP at each visit.

OTHER OUTCOMES:
safety of angle intervention surgeries | 1 months
  The main observation includes recording intraoperative and postoperative complications, including hyphema, choroidal detachment, cyclodialysis, persistent hypotony, corneal decompensation, and intraocular inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Xinbo Gao, MD, Principal Investigator — State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan ophthalmic center, Guangzhou, Guangdong, China